CLINICAL TRIAL: NCT00522587
Title: Sevoflurane-Remifentanil Interaction: Multiple Response Surfaces, Validation of Calibration Stimuli, Validation of the Intraoperative Isobole Concept and Investigating Remifentanil Induced Opioid Tolerance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007/242
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (12):
- 1 (Experimental): Fixed sevoflurane dose 1
  Interventions: Drug: Fixed sevoflurane dose 1
- 2 (Experimental): Fixed sevoflurane dose 2
  Interventions: Drug: Fixed sevoflurane dose 2
- 3 (Experimental): Fixed sevoflurane dose 3
  Interventions: Drug: Fixed sevoflurane dose 3
- 4 (Experimental): Fixed sevoflurane dose 4
  Interventions: Drug: Fixed sevoflurane dose 4
- 5 (Experimental): Fixed sevoflurane dose 5
  Interventions: Drug: Fixed sevoflurane dose 5
- 6 (Experimental): Fixed sevoflurane dose 6
  Interventions: Drug: Fixed sevoflurane dose 6
- 7 (Experimental): Fixed remifentanil dose 1
  Interventions: Drug: Fixed remifentanil dose 1
- 8 (Experimental): Fixed remifentanil dose 2
  Interventions: Drug: Fixed remifentanil dose 2
- 9 (Experimental): Fixed remifentanil dose 3
  Interventions: Drug: Fixed remifentanil dose 3
- 10 (Experimental): Fixed remifentanil dose 4
  Interventions: Drug: Fixed remifentanil dose 4
- 11 (Experimental): Fixed remifentanil dose 5
  Interventions: Drug: Fixed remifentanil dose 5
- 12 (Experimental): Fixed remifentanil dose 6
  Interventions: Drug: Fixed remifentanil dose 6

INTERVENTIONS:
Drug: Fixed sevoflurane dose 1 — Dose 1 of sevoflurane
  Arms: 1
Drug: Fixed sevoflurane dose 2 — Dose 2 of sevoflurane
  Arms: 2
Drug: Fixed sevoflurane dose 3 — Dose 3 of sevoflurane
  Arms: 3
Drug: Fixed sevoflurane dose 4 — Dose 4 of sevoflurane
  Arms: 4
Drug: Fixed sevoflurane dose 5 — Dose 5 of sevoflurane
  Arms: 5
Drug: Fixed sevoflurane dose 6 — Dose 6 of sevoflurane
  Arms: 6
Drug: Fixed remifentanil dose 1 — Dose 1 of remifentanil
  Arms: 7
Drug: Fixed remifentanil dose 2 — Dose 2 of remifentanil
  Arms: 8
Drug: Fixed remifentanil dose 3 — Dose 3 of remifentanil
  Arms: 9
Drug: Fixed remifentanil dose 4 — Dose 4 of remifentanil
  Arms: 10
Drug: Fixed remifentanil dose 5 — Dose 5 of remifentanil
  Arms: 11
Drug: Fixed remifentanil dose 6 — Dose 6 of remifentanil
  Arms: 12

SUMMARY:
During this study, the pharmacodynamic interactions between sevoflurane and remifentanil will be studied.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesia class I and II patients
* Aged 18-60 years
* Scheduled for surgery under general anesthesia

Exclusion Criteria:

* Weight less than 70% or more than 130% of ideal body weight
* Neurological disorder
* Diseases involving the cardiovascular system (hypertension, coronary artery disease, prior acute myocardial infarction (AMI), any valvular and/or muscular disease involving decrease of the ejection fraction, arrhythmias, which are either symptomatic or require continuous medication/pacemaker/automatic implantable cardioverter defibrillator [AICD])
* Pulmonary disease including asthma, severe chronic obstructive pulmonary disease (COPD), etc.
* Gastric diseases including reflux, endocrinological diseases
* Recent use of psycho-active medication, including alcohol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-04; Primary Completion 2009-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
EEG depression and arousal reactions in response to different clinically relevant stimuli | 60 to 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Michel Struys, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be